CLINICAL TRIAL: NCT03698864
Title: An Open-Label Study to Evaluate the Safety and Tolerability of PCS499 for the Treatment of Necrobiosis Lipoidica
Brief Title: A Study to Evaluate the Safety and Tolerability of PCS499 for the Treatment of Necrobiosis Lipoidica
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Processa Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCS499-NL01
Record Dates: First submitted 2018-10-01; First posted 2018-10-09 (Actual); Results first posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Necrobiosis Lipoidica
MeSH Terms: conditions — Necrobiosis Lipoidica

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PCS499 900mg twice a day (Experimental)
  Interventions: Drug: PCS499

INTERVENTIONS:
Drug: PCS499 — PCS499 900mg twice a day with food

SUMMARY:
This is an open-label study that will evaluate the safety of PCS499 for the treatment of necrobiosis lipoidica (NL) and will inform the design of future studies. Approximately 12 NL patients (6-9 patients without ulceration and 3-6 patients with ulceration) who also meet other inclusion/exclusion criteria will be enrolled in the study. The primary objective of this study is to evaluate the safety and tolerability profile of PCS499 in patients with Necrobiosis Lipoidica.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients age 18 to 80 years of age, inclusive, at Screening.
2. Biopsy-confirmed diagnosis of NL. Biopsies of continually active lesions performed outside of this clinical study will need to be reviewed and the diagnosis confirmed by the study pathologist. For patients with no previous history of biopsy, no biopsy within the previous 5 years, a biopsy that is not confirmed to be NL, or newly active lesion, a biopsy to confirm a diagnosis of NL will be performed at the Screening visit.
3. Reference NL lesion with a score of 2 or greater on the Investigator Global Assessment: Necrobiosis Lipoidica (IGA:NL) Activity scale AND surface area with minimum size of 10 cm2. If more than one lesion is present, the reference lesion area is the lesion with the highest disease severity.
4. Women of childbearing potential must have a negative serum pregnancy test at the Screening Visit and a negative urine pregnancy test at Baseline before dosing.
5. Women of childbearing potential must use one of the following acceptable methods of contraception throughout the study: oral contraceptive medication, intrauterine device (IUD), hormonal implants, injectable contraceptive medications, double-barrier methods, or tubal ligation.
6. Females who are postmenopausal (age-related amenorrhea >= 12 consecutive months and increased follicle-stimulating hormone [FSH] > 40 mIU/mL. If necessary to confirm postmenopausal status, an FSH will be drawn at Screening) or who have undergone hysterectomy or bilateral oophorectomy are exempt from pregnancy testing.
7. Male patients must be willing to use appropriate contraceptive measures and refrain from sexual activity with any female who is pregnant or lactating.
8. Patient must be willing and able to swallow whole tablets.
9. Patient must be willing and able to comply with study procedures.
10. Patient must be willing and able to provide signed, informed consent.

Exclusion Criteria:

1. Current or previous (within 4 weeks of Baseline) treatment with:

   1. Oral, topical, or intralesional corticosteroids;
   2. Systemic pentoxifylline, theophylline, or cilostazol
   3. Oral or topical retinoid;
   4. Other systemic or topical immunosuppressant drugs, including but not limited to calcineurin inhibitors (e.g., tacrolimus), thalidomide, apremilast, anti-malarials (e.g., hydroxychloroquine, chloroquine), cyclosporine, mycophenolate mofetil, azathioprine, methotrexate, etc.
2. Current or previous (within 12 weeks of Baseline) treatment with any biologic therapy (e.g., adalimumab, etanercept, infliximab, anakinra, etc.).
3. Phototherapy/photochemotherapy (NBUVB, UVB, PUVA) within 6 weeks prior to Baseline
4. Skin grafting, or other surgical procedure (other than debridement) within 6 weeks prior to Baseline.
5. History of drug allergy, including but not limited to pentoxifylline or other xanthine derivatives, or other allergy, which in the opinion of the Investigator, contraindicates participation.
6. Anticipated concurrent use of a strong CYP1A2 inhibiting drug, including but not limited to cimetidine and/or fluvoxamine, during the course of the study (after Screening).
7. Fever (>38°C), or chronic, persistent, or recurring infection(s) at Screening or Baseline.
8. Any infection requiring oral antimicrobial therapy within 2 weeks prior to Baseline or any infection requiring parenteral antibiotics or hospitalization within 12 weeks prior to Baseline. Any treatment for such infections must have been completed and the infection cured for at least 2 weeks prior to Baseline.
9. History of sarcoidosis, pyoderma gangrenosum, or any other disorder (in the judgment of the Investigator) that would interfere with the evaluation of NL or require protocol prohibited medication.
10. History of any life threatening infection or sepsis within 12 months of Baseline:
11. Clinically significant cardiac disease including but not limited to unstable angina, acute myocardial infarction within 6 months of Baseline, and arrhythmia requiring therapy.
12. Patient has QTc interval ≥ 480 milliseconds on Screening Electrocardiogram (ECG); a second Screening ECG may be done at investigator's discretion but the average of the two QTc screening intervals must not be ≥ 480 milliseconds.History of cerebral hemorrhage, cerebrovascular accident, transient ischemic attack, gastrointestinal bleeding, or retinal hemorrhage within 6 months of Baseline.
13. History of cerebral hemorrhage, cerebrovascular accident, transient ischemic attack, gastrointestinal bleeding, or retinal hemorrhage within 6 months of Baseline.
14. Patient has active or history of neoplastic disease (except for adequately treated non-invasive basal cell and/or squamous cell carcinoma or carcinoma in situ of the cervix) within the past 5 years prior to Baseline.
15. Presence of clinically significant medical condition(s) including but not limited to: renal, hepatic, cardiovascular, hematological, gastrointestinal, endocrine, pulmonary, neurological, psychiatric, substance abuse, and/or any other clinically significant disease or disorder, which in the opinion of the Investigator (by its nature or by being inadequately controlled), may put the patient at risk due to participation in the study, influence the results of the study, and/or affect the patient's ability to complete the study.
16. History of or current diagnosis of active tuberculosis (TB); undergoing treatment for latent TB infection (LTBI); untreated LTBI (as determined by documented results within 3 months of the Screening Visit of a positive TB skin test with purified protein derivative with induration >= 5 millimeter (mm), or a positive QuantiFERON-TB test or positive or borderline T-Spot [Elispot] test); or positive TB test at Screening. Subjects with documented completion of appropriate LTBI treatment would not be excluded and are not required to be tested.
17. Vaccination with live or live-attenuated virus vaccine within 1 month prior to Baseline.
18. The results of the following laboratory tests performed at the central laboratory at Screening meet any of the criteria below:

    1. Hemoglobin < 8.0 g/dL (International System of Units (SI): < 80 g/L);
    2. White blood cells < 3.0 x 10^3 cells/mm^3 (SI: < 3.0 x 10^9 cells/L);
    3. Neutrophils < 1.0 x 10^3 cells/mm^3 (SI: < 1.0 x 10^9 cells/L);
    4. Lymphocytes < 0.5 x 10^3 cells/mm^3 (SI: < 0.5 x 10^9 cells/L);
    5. Platelets < 100 x 10^3 cells/mm^3 (SI: < 100 x 10^9 cells/L)
    6. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and/or alkaline phosphatase (ALP) ≥ 2 x upper limit of normal (ULN);
    7. Total bilirubin level ≥ 2 x ULN unless the individual has been diagnosed with Gilbert's disease and this is clearly documented;
    8. Estimated glomerular filtration rate < 40 mL/min/1.73 m^2 based on the Modification of Diet in Renal Disease (MDRD) formula.
    9. Positive HIV serology
    10. Evidence of active Hepatitis B Virus (HBV) infection
    11. Evidence of active Hepatitis C Virus (HCV) infection
19. Women who are pregnant or breastfeeding.
20. Patient unwilling or unable to swallow tablets whole.
21. Any other medical condition, serious intercurrent illness, or extenuating circumstance that, in the opinion of the Investigator, would preclude participation in the study.
22. Use of any investigational product within 30 days prior to Baseline or currently enrolled in another study that involves clinical investigations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maya Das, MD, Study Director — Processa Pharmaceuticals
Locations (2):
- United States (2):
  - Processa Investigational Site, Philadelphia, Pennsylvania
  - Processa Investigational Site, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PCS499 900mg Twice a Day
Started | 12
Completed | 10
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: ulcerated (2 of 12) non-ulcerated (10 of 12)
Arm/Group | PCS499 900mg Twice a Day
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (13.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Screening Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 28.80 (3.338)
Number of Days since NL diagnosis to screening [Mean (Standard Deviation); unit: days] | 4498.25 (3759.580)

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Patients With Adverse Events
Description: Evaluation of Adverse Events/Serious Adverse Events (by type, severity, and relatedness)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | PCS499 900mg Twice a Day
Number analyzed (Participants) | 12
Participants | 10

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | PCS499 900mg Twice a Day
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 10/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PCS499 900mg Twice a Day (N=12)
Nausea (Gastrointestinal disorders) | 4
Abdominal Discomfort (Gastrointestinal disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 1
Influenza (Infections and infestations) | 2
Anaemia (Blood and lymphatic system disorders) | 1
Ulcer (General disorders) | 1
Abcess (Infections and infestations) | 1
Gastroenteritis Viral (Infections and infestations) | 1
Rash Pustular (Infections and infestations) | 1
Tooth Abcess (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1
Eschar (Injury, poisoning and procedural complications) | 1
Blood Glucose Increased (Investigations) | 1
Electrocardiogram Qt Prolonged (Investigations) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
open label study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT03698864/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/64/NCT03698864/SAP_001.pdf